CLINICAL TRIAL: NCT01981915
Title: Optimum Insufflation Capacity and Peak Cough Flow Augmentation in Patients With Neuromuscular Disease
Brief Title: Optimum Insufflation Capacity in NMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universität Duisburg-Essen (Other)
Collaborators: Weinmann Geräte für Medizin GmbH + Co. KG (Industry)
Responsible Party: Principal Investigator, Uwe Mellies, Priv.-Doz. Dr. med., Universität Duisburg-Essen
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: OIC2013
Record Dates: First submitted 2013-10-11; First posted 2013-11-13 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Duchenne Muscular Dystrophy; Spinal Muscular Atrophy; Chronic Respiratory Insufficiency
Keywords: Cough augmentation; Peak cough flow; hyperinsufflation
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Muscular Atrophy, Spinal | interventions — Intermittent Positive-Pressure Breathing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lung Insufflation Volume (Experimental): Measurement of the lung volume after hyperinsufflation with positive pressure by IPPB or LIAM
  Interventions: Procedure: IPPB; Procedure: LIAM
- Peak Cough Flow (Experimental): Measurement of the peak cough flow after hyperinsufflation with positive pressure by IPPB or LIAM
  Interventions: Procedure: IPPB; Procedure: LIAM

INTERVENTIONS:
Procedure: IPPB — Lung insufflation with positive pressure using IPPB up from 10 to 40 mbar in 5 mbar increments and consecutive measurement of the insufflation volume
  Other Names: Intermittent Positive Pressure Breathing = IPPB
Procedure: LIAM — Lung insufflation using the Lung Insufflation Assist maneuver of the Ventilogic LS mechanical ventilator (Weinmann Germany) with positive pressure up from 10 to 40 mbar in 5 mbar increments and consecutive measurement of the insufflation volume
  Other Names: LIAM = Lung Insufflation Assist Maneuver

SUMMARY:
Patients with underlying neuromuscular disorder (NMD) often suffer from weakness in the inspiratory and expiratory muscles. Consequently they do not have the strength to generate the minimum flow of 160 to 300 liters/minute for an efficient cough function. The restricted cough function allows secretion to accumulate, which in turn causes narrowing of the airway lumen and makes ventilation of the neuromuscular patient even more difficult. The patient's susceptibility to infection increases again and the vicious circle repeats itself. Severe secretion retention may even lead to ventilator failure. Effective secretion and cough management instead reduces the risk for stay in hospital. Therefore, secretion and cough management is a mandatory part of the therapeutic concept for treating patients with neuromuscular disease.

The therapeutic efficacy of the Lung Insufflation Assist Maneuver(LIA) integrated in the ventilator VENTIlogic LS-plus manufactured by Weinmann GmbH+Co KG was studied in a pilot study carried out by the Dep. for Pediatric Pulmonology and Sleep Medicine at the University Hospital of Essen/Germany in cooperation with Research & Development at Weinmann GmbH &Co KG, Germany . The objective of the pilot study was to examine the therapeutic efficacy of LIAM as a cough support function in patients with neuromuscular disease and indications for mechanical ventilation.

We hypothesized that i) a certain insufflation maneuver pressure may be optimal to achieve the highest individual peak cough flow and ii) that this pressure is below the pressure needed to achieve the maximum insufflation capacity. We define the lowest insufflation capacity at which the best individual PCF can be achieved as optimum insufflation capacity (OIC). The study was performed using two different techniques in order to demonstrate that findings are not dependent on maneuver details but are rather based on effects of maneuver pressure. The protocol was limited to techniques which do not require breath stacking: i) insufflation with an Intermittend Positive Pressure (IPPB) device and ii) with the VENTIlogic LS using LIAM.

ELIGIBILITY:
Inclusion Criteria:

* neuromuscular disorder
* respiratory insufficiency
* use of home mechanical ventilation

Exclusion Criteria:

* acute illness
* history of pneumothorax

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
insufflation capacity | change of lung volume with the procedure; during hospital stay on average 3 days
  Lung volume was measured during spontaneous breathing and after a lung insufflation assist maneuver.

SECONDARY OUTCOMES:
Peak cough flow | change of peak cough flow with the procedure; during hospital stay on average 3 days
  Peak cough flow was measured during spontaneous breathing and after a lung insufflation assist maneuver.

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Mellies, MD, Principal Investigator — University of Essen, Germany
Locations (1):
- University of Essen, Children's Hospital, Dep. of Pediatric Pulmonology, Essen, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Dohna-Schwake C, Ragette R, Teschler H, Voit T, Mellies U. Predictors of severe chest infections in pediatric neuromuscular disorders. Neuromuscul Disord. 2006 May;16(5):325-8. doi: 10.1016/j.nmd.2006.02.003. Epub 2006 Apr 18. PMID 16621559
- [Background] Ishikawa Y, Bach JR, Komaroff E, Miura T, Jackson-Parekh R. Cough augmentation in Duchenne muscular dystrophy. Am J Phys Med Rehabil. 2008 Sep;87(9):726-30. doi: 10.1097/PHM.0b013e31817f99a8. PMID 18716484
- [Background] Bach JR, Mahajan K, Lipa B, Saporito L, Goncalves M, Komaroff E. Lung insufflation capacity in neuromuscular disease. Am J Phys Med Rehabil. 2008 Sep;87(9):720-5. doi: 10.1097/PHM.0b013e31817fb26f. PMID 18716483
- [Background] Hahneberger RW. Applanation tonometry in the conscious cynomolgus monkey (Macaca fascicularis). Acta Ophthalmol (Copenh). 1976 Jul;54(3):311-9. doi: 10.1111/j.1755-3768.1976.tb01260.x. PMID 821306